CLINICAL TRIAL: NCT06396689
Title: NapBiome: Targeting Gut Microbiota and Sleep Rhythm to Improve Developmental and Behavioral Outcomes in Early Childhood
Acronym: NapBiome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Petra Zimmermann (Other)
Collaborators: University of Luzern (Other); Swiss Federal Institute of Technology in Zurich (ETHZ) (Unknown)
Responsible Party: Sponsor-Investigator, Petra Zimmermann, Deputy Head of Paediatrics, Head of Paediatric Infectious Diseases, University of Fribourg
Organization: University of Fribourg (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 123
Record Dates: First submitted 2024-04-10; First posted 2024-05-02 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Sleep Problem; Neurobehavioral Manifestations
Keywords: microbiome; infant; gut; metagenomics; development; metabolics; pre-term; probiotics; synbiotics; brain-gut
MeSH Terms: conditions — Parasomnias; Neurobehavioral Manifestations; Premature Birth | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Preterm-born infants assigned to "synbiotics" (PRET-SYN) (Active Comparator)
  Interventions: Dietary Supplement: Synbiotic
- Preterm-born infants to "placebo" (PRET-PLC) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Term-born infants to "synbiotics" (TERM-SYN) (Active Comparator)
  Interventions: Dietary Supplement: Synbiotic
- Term-born infants to "placebo" (TERM-PLC) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — The capsule contains Lactobacillus helveticus R0052, Bifidobacterium infantis R0033, and Bifidobacterium bifidum R0071 (3 billion bacteria per capsule), as well as zinc oxide, potato starch fructooligosaccharides, coating agent, methyl hydroxypropyl cellulose, anti-caking agent and magnesium stearat
  Arms: Preterm-born infants assigned to "synbiotics" (PRET-SYN); Term-born infants to "synbiotics" (TERM-SYN)
Dietary Supplement: Placebo — The capsule contains zinc oxide, coating agent, methyl hydroxypropyl cellulose, anti-caking agent and magnesium stearat
  Arms: Preterm-born infants to "placebo" (PRET-PLC); Term-born infants to "placebo" (TERM-PLC)

SUMMARY:
The gut-brain axis plays a crucial role in the regulation and development of psychological and physical processes. The first year of life is a critical period for the development of the gut microbiome, which parallels important milestones in establishing sleep rhythm and neurodevelopment. Growing evidence suggests that the gut microbiome influences sleep, cognition, and early neurodevelopment. For term and preterm-born infants, difficulties in sleep regulation can have major consequences on infants' health, attachment between infants and their caregivers, and can even lead to life-threatening consequences such as shaken-baby syndrome. Preterm born infants are at even higher risk for sleep and neurodevelopmental problems. Although neonatal care has improved over recent decades, preterm birth rates continue to rise and lead to a wide range of neurodevelopmental disabilities that are unaddressed with current therapies. Given the importance of sleep and the gut microbiome for brain maturation, neurodevelopment, and behavior, identifying effective interventions within the gut-brain axis at the beginning of life is likely to have long-term implications for health and development of at-risk infants.

The aims of this project are to I) demonstrate the association between the gut microbiome, sleep patterns and health outcomes in children up to two years of age; and II) to leverage gut microbiome-brain-sleep interactions to develop new intervention strategies for at-risk infants. The investigators hypothesize that the establishment of a healthy gut microbiome during early life is crucial for both short- and long-term child health outcomes, as dysbiosis can harm sleep regulation, brain maturation, and neurobehavioral development. The investigators predict that the administration of synbiotics improves microbiota establishment, sleep rhythm, and neurodevelopmental outcomes.

This project integrates a randomized controlled trial (RCT), ex vivo, and in silico experiments with I) key technology platforms for computational modeling to capture the ontogenic norms of gut microbiota; II) neuronal and actimetry-based quantification of multidimensional aspects of infant sleep; III) breath metabolomics (exhalomics) of host and microbiome metabolism; and IV) high-throughput ex vivo models for investigating host-microbiome interactions. Outcomes include I) an understanding of age-normative microbiome composition, its variation (circadian, inter-individual), and the factors that influence the microbiome's plasticity throughout infancy; II) actionable knowledge of microbial species and metabolism that can be targeted to modify sleep regulation and improve neurodevelopmental outcomes, especially in at-risk infants (e.g., preterm-born); III) microbial and metabolic biomarkers with diagnostic potential for later regulatory and behavioral problems; and IV) an open-source analytical "toolbox" for microbial multi-omics that can be immediately applied in other areas of microbiome-host research. To achieve these goals, our strategy combines multiple disciplines focusing on factors that exert the greatest influence on health during infancy: the gut microbiome, sleep regulation, and neurodevelopment.

The impact of this project is substantial and globally relevant, as it advances possible treatment options for supporting neurodevelopmental health in preterm- and term-born infants, explores novel translational approaches for addressing regulatory difficulties, and provides key information for tailored prophylactic synbiotics and possible development of "post-biotics". Further, the study supports the investigation of biomarkers for neurodevelopment and advances early prevention of developmental and mental illnesses.

ELIGIBILITY:
Inclusion Criteria:

Preterm-arm:

* neonates born between a gestational age of 34 0/7 to 36 6/7 weeks
* partially breast-fed at the time of inclusion

Term-arm

* neonates born at a gestational age of ≥ 37 0/7 weeks Infants need to be
* partially breast-fed at the time of inclusion

Exclusion Criteria:

Infants who

* receive probiotics outside the trial design
* have a birth weight < 1500 g
* were prenatally drug-exposed (cannabis, cocaine, heroin, opiates, and alcohol)
* have suspected or confirmed immunodeficiency
* have an underlying disease (excluding transient conditions such as alimentation problems, hyperbilirubinemia, hypoglycaemia, anemia, respiratory distress syndrome or apnea-bradycardia syndrome), congenital malformations, central nervous system disease or injury or congenital infections

Ages: 0 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Sleep-wake behavior | up to two years of age
  Brief Infant Sleep Questionnaire BISQ, actinometry and sleep-wake diary
Neuronal connectivity | up to two years of age
  High-density EEG during sleep
Neurobehavioral development | up to two years of age
  Bayley Scales of Infant Development
Behavior | up to two years of age
  Infant Behavior Questionnaire
Gut microbiota | up to two years of age
  Composition of stool microbiota
Stool metabolome | up to two years of age
  Composition of stool metabolites
Breath metabolome | up to two years of age
  Composition of breath metabolites

SECONDARY OUTCOMES:
Eczema | up to two years of age
  SCORing Atopic Dermatitis scoring system (SCORAD)
Food allergy | up to two years of age
  Skin prick test
Rates of infection | up to two years of age
  Number of episodes
Breast milk microbiota | up to two years of age
  Composition investigated trough shotgun metagenomic sequencing
Nasal microbiota | up to two years of age
  Composition investigated trough shotgun metagenomic sequencing
Oral microbiota | up to two years of age
  Composition investigated trough shotgun metagenomic sequencing

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Hopital cantonal Fribourg, Fribourg, Canton of Fribourg
  - Cantonal Hospital, Lucerne, Canton of Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zimmermann P, Kurth S, Giannoukos S, Stocker M, Bokulich NA. NapBiome trial: Targeting gut microbiota to improve sleep rhythm and developmental and behavioural outcomes in early childhood in a birth cohort in Switzerland - a study protocol. BMJ Open. 2025 Mar 3;15(3):e092938. doi: 10.1136/bmjopen-2024-092938. PMID 40032396